CLINICAL TRIAL: NCT05882864
Title: Efficacy of Ginger Muco-bioadhesive Gel in Management of Oral Lichen Planus: A Randomized Controlled Clinical Trial With Immunohistochemical Analysis
Brief Title: Efficacy of Ginger Muco-bioadhesive Gel in Management of Oral Lichen Planus With Immunohistochemical Analysis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Herbs in oral medicine
Record Dates: First submitted 2023-05-22; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Oral Lichen Planus
MeSH Terms: conditions — Lichen Planus, Oral | interventions — gingerol; Triamcinolone Acetonide

STUDY DESIGN:
Intervention Model Description: Group I Will include 14 patients receiving topical ginger extract 1% four times per day (after every meal and before going to bed) for eight weeks (Zakaria et al., 2020).
  Group II Will include 14 patients receiving topical steroid (triamcinolone acetonide 0.1%) four times per day for eight weeks (Laeijendecker et al., 2006)
Who Masked: Participant, Care Provider
Masking Description: The study is designed to be a prospective randomized double blind 2 parallel arms controlled clinical trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topical 6-Gingerol Group (Active Comparator): Group I Will include 14 patients receiving topical ginger extract 1% four times per day (after every meal and before going to bed) for eight weeks (Zakaria et al., 2020).
  Interventions: Drug: 6-Gingerol
- Topical Steroid Group (Active Comparator): Group II Will include 14 patients receiving topical steroid (triamcinolone acetonide 0.1%) four times per day for eight weeks (Laeijendecker et al., 2006)
  In the fourth and eighth weeks, topical anti-fungal will be applied by a third-party medical personnel to avoid 2ry candidiasis for this group.
  Interventions: Drug: Triamcinolone Acetonide 0.1% Oromucosal Paste

INTERVENTIONS:
Drug: 6-Gingerol — 6-gingerol gel will be applied locally to the participants suffering from oral lichen planus
  Arms: Topical 6-Gingerol Group
Drug: Triamcinolone Acetonide 0.1% Oromucosal Paste — Triamcinolone Acetonide 0.1% gel will be applied locally to the participants suffering from oral lichen planus
  Arms: Topical Steroid Group

SUMMARY:
1. Compare the clinical efficacy of topical ginger extract versus triamcinolone acetonide 0.1% for symptomatic oral lichen planus (Primary Objective).
2. Investigate using immunohistochemical analysis the effect of the two different treatment modalities on FasL expression in oral lichen planus lesions (Secondary Objective).

ELIGIBILITY:
Inclusion Criteria:

* Males or females, aged from 40 to 60 years.
* Clinically proven painful Bullous/erosive (score 4) or atrophic (score 3) forms of OLP confirmed by the presence of red or erythromatous changes, or shallow ulcerations with fine lacy lines at the periphery of the lesion accentuated by stretching and not eliminated by rubbing (Wickham's striae) (Lozada-Nur and Miranda, 1997)
* Histopathologically, proven Bullous/erosive (score 4) or atrophic (score 3) forms of OLP confirmed by the presence of accepted histopathological criteria for lichen planus; basal cell liquefaction, band like lymphocytic infiltrate at the epithelial-stromal junction with degeneration of basal cell region (Ellis, 1967; Van der Meij and Van der Waal, 2003).

Exclusion Criteria:

* History of drug induced lichenoid lesions.
* Presence of systemic conditions as; serious active or recurrent infections, malignancy, diabetes mellitus, hypertension, or significant heart, liver, or renal diseases. Assessed using medical questionnaire guided by Cornell Medical Index (Pendleton et al., 2004).
* Smoking.
* Known hypersensitivity or severe adverse effects to the treatment drugs or to any ingredient of their preparation as mentioned in medical history.
* Pregnancy or breast-feeding.
* History of previous treatments potentially effective on OLP such as antimalarial agents, retinoids, corticosteroids or immunosuppressive drugs from less than 2 weeks for topical medications, and 4 weeks for systemic medications prior to starting the study (Swift et al., 2005).
* Patients suffering from lichen planus skin lesions.
* Loss of pliability or flexibility in the tissues involved by the oral lesions of lichen planus.
* Histological signs of epithelial dysplasia or lichenoid lesions within the biopsied.
* Refusing to participate in the study.
* Vulnerable groups (handicapped, orphans and prisoners).

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Ginger Muco-bioadhesive Gel in Management of Oral Lichen Planus | Baseline
  Analysis of 6-Gingerol gel in Management of Oral Lichen Plauns using Immunohistochemistry

REFERENCES:
- [Background] Ahn SI, Lee JK, Youn HS. Inhibition of homodimerization of toll-like receptor 4 by 6-shogaol. Mol Cells. 2009 Feb 28;27(2):211-5. doi: 10.1007/s10059-009-0026-y. Epub 2009 Feb 20. PMID 19277504
- [Background] Ali BH, Blunden G, Tanira MO, Nemmar A. Some phytochemical, pharmacological and toxicological properties of ginger (Zingiber officinale Roscoe): a review of recent research. Food Chem Toxicol. 2008 Feb;46(2):409-20. doi: 10.1016/j.fct.2007.09.085. Epub 2007 Sep 18. PMID 17950516
- [Background] Anitua E, Pinas L, Alkhraisat MH. Histopathological features of oral lichen planus and its response to corticosteroid therapy: A retrospective study. Medicine (Baltimore). 2019 Dec;98(51):e18321. doi: 10.1097/MD.0000000000018321. PMID 31860983
- [Background] Canto AM, Muller H, Freitas RR, Santos PS. Oral lichen planus (OLP): clinical and complementary diagnosis. An Bras Dermatol. 2010 Sep-Oct;85(5):669-75. doi: 10.1590/s0365-05962010000500010. PMID 21152791
- [Background] Chainani-Wu N, Silverman S Jr, Lozada-Nur F, Mayer P, Watson JJ. Oral lichen planus: patient profile, disease progression and treatment responses. J Am Dent Assoc. 2001 Jul;132(7):901-9. doi: 10.14219/jada.archive.2001.0302. PMID 11480643
- [Background] Cheng A, Mann C. Oral erosive lichen planus treated with efalizumab. Arch Dermatol. 2006 Jun;142(6):680-2. doi: 10.1001/archderm.142.6.680. No abstract available. PMID 16785369
- [Background] Choonhakarn C, Busaracome P, Sripanidkulchai B, Sarakarn P. The efficacy of aloe vera gel in the treatment of oral lichen planus: a randomized controlled trial. Br J Dermatol. 2008 Mar;158(3):573-7. doi: 10.1111/j.1365-2133.2007.08370.x. Epub 2007 Dec 17. PMID 18093246
- [Background] Dragovich T, Rudin CM, Thompson CB. Signal transduction pathways that regulate cell survival and cell death. Oncogene. 1998 Dec 24;17(25):3207-13. doi: 10.1038/sj.onc.1202587. PMID 9916983
- [Background] Eisenberg E. Oral lichen planus: a benign lesion. J Oral Maxillofac Surg. 2000 Nov;58(11):1278-85. doi: 10.1053/joms.2000.16629. No abstract available. PMID 11078140
- [Background] Ellis FA. Histopathology of lichen planus based on analysis of one hundred biopsy specimens. J Invest Dermatol. 1967 Feb;48(2):143-8. doi: 10.1038/jid.1967.23. No abstract available. PMID 6020677
- [Background] Eversole LR. Immunopathogenesis of oral lichen planus and recurrent aphthous stomatitis. Semin Cutan Med Surg. 1997 Dec;16(4):284-94. doi: 10.1016/s1085-5629(97)80018-1. PMID 9421220
- [Background] Farhi D, Dupin N. Pathophysiology, etiologic factors, and clinical management of oral lichen planus, part I: facts and controversies. Clin Dermatol. 2010 Jan-Feb;28(1):100-8. doi: 10.1016/j.clindermatol.2009.03.004. PMID 20082959
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Gonzalez-Moles MA, Warnakulasuriya S, Gonzalez-Ruiz I, Gonzalez-Ruiz L, Ayen A, Lenouvel D, Ruiz-Avila I, Ramos-Garcia P. Worldwide prevalence of oral lichen planus: A systematic review and meta-analysis. Oral Dis. 2021 May;27(4):813-828. doi: 10.1111/odi.13323. Epub 2020 Apr 2. PMID 32144836
- [Background] Gorouhi F, Davari P, Fazel N. Cutaneous and mucosal lichen planus: a comprehensive review of clinical subtypes, risk factors, diagnosis, and prognosis. ScientificWorldJournal. 2014 Jan 30;2014:742826. doi: 10.1155/2014/742826. eCollection 2014. PMID 24672362
- [Background] Grzanna R, Lindmark L, Frondoza CG. Ginger--an herbal medicinal product with broad anti-inflammatory actions. J Med Food. 2005 Summer;8(2):125-32. doi: 10.1089/jmf.2005.8.125. PMID 16117603
- [Background] Haghpanah P, Moghadamnia AA, Zarghami A, Motallebnejad M. Muco-bioadhesive containing ginger officinal e extract in the management of recurrent aphthous stomatitis: A randomized clinical study. Caspian J Intern Med. 2015 Winter;6(1):3-8. PMID 26221489
- [Background] Ismail SB, Kumar SK, Zain RB. Oral lichen planus and lichenoid reactions: etiopathogenesis, diagnosis, management and malignant transformation. J Oral Sci. 2007 Jun;49(2):89-106. doi: 10.2334/josnusd.49.89. PMID 17634721
- [Background] Jolad SD, Lantz RC, Solyom AM, Chen GJ, Bates RB, Timmermann BN. Fresh organically grown ginger (Zingiber officinale): composition and effects on LPS-induced PGE2 production. Phytochemistry. 2004 Jul;65(13):1937-54. doi: 10.1016/j.phytochem.2004.06.008. PMID 15280001
- [Background] Laeijendecker R, Tank B, Dekker SK, Neumann HA. A comparison of treatment of oral lichen planus with topical tacrolimus and triamcinolone acetonide ointment. Acta Derm Venereol. 2006;86(3):227-9. doi: 10.2340/00015555-0070. PMID 16710580
- [Background] Li C, Tang X, Zheng X, Ge S, Wen H, Lin X, Chen Z, Lu L. Global Prevalence and Incidence Estimates of Oral Lichen Planus: A Systematic Review and Meta-analysis. JAMA Dermatol. 2020 Feb 1;156(2):172-181. doi: 10.1001/jamadermatol.2019.3797. PMID 31895418
- [Background] Lopez-Jornet P, Camacho-Alonso F, Salazar-Sanchez N. Topical tacrolimus and pimecrolimus in the treatment of oral lichen planus: an update. J Oral Pathol Med. 2010 Mar;39(3):201-5. doi: 10.1111/j.1600-0714.2009.00830.x. Epub 2009 Nov 20. PMID 19943858
- [Background] Lozada-Nur F, Miranda C. Oral lichen planus: epidemiology, clinical characteristics, and associated diseases. Semin Cutan Med Surg. 1997 Dec;16(4):273-7. doi: 10.1016/s1085-5629(97)80016-8. PMID 9421218
- [Background] Mashhadi NS, Ghiasvand R, Askari G, Feizi A, Hariri M, Darvishi L, Barani A, Taghiyar M, Shiranian A, Hajishafiee M. Influence of ginger and cinnamon intake on inflammation and muscle soreness endued by exercise in Iranian female athletes. Int J Prev Med. 2013 Apr;4(Suppl 1):S11-5. PMID 23717759
- [Background] Mozaffari HR, Sharifi R, Sadeghi M. Prevalence of Oral Lichen Planus in Diabetes Mellitus: a Meta-Analysis Study. Acta Inform Med. 2016 Dec;24(6):390-393. doi: 10.5455/aim.2016.24.390-393. PMID 28077900
- [Background] Nagata S. Apoptosis regulated by a death factor and its receptor: Fas ligand and Fas. Philos Trans R Soc Lond B Biol Sci. 1994 Aug 30;345(1313):281-7. doi: 10.1098/rstb.1994.0107. PMID 7531345
- [Background] Nagata S. Fas ligand-induced apoptosis. Annu Rev Genet. 1999;33:29-55. doi: 10.1146/annurev.genet.33.1.29. PMID 10690403
- [Background] Pedersen A. Abnormal EBV immune status in oral lichen planus. Oral Dis. 1996 Jun;2(2):125-8. doi: 10.1111/j.1601-0825.1996.tb00212.x. PMID 8957924
- [Background] Pendleton N, Clague JE, Horan MA, Rabbitt PM, Jones M, Coward R, Lowe C, McInnes L. Concordance of Cornell medical index self-reports to structured clinical assessment for the identification of physical health status. Arch Gerontol Geriatr. 2004 May-Jun;38(3):261-9. doi: 10.1016/j.archger.2003.10.005. PMID 15066312
- [Background] Peter ME, Krammer PH. Mechanisms of CD95 (APO-1/Fas)-mediated apoptosis. Curr Opin Immunol. 1998 Oct;10(5):545-51. doi: 10.1016/s0952-7915(98)80222-7. PMID 9794832
- [Background] Prasad S, Tyagi AK. Ginger and its constituents: role in prevention and treatment of gastrointestinal cancer. Gastroenterol Res Pract. 2015;2015:142979. doi: 10.1155/2015/142979. Epub 2015 Mar 8. PMID 25838819
- [Background] Radwan-Oczko M, Zwyrtek E, Owczarek JE, Szczesniak D. Psychopathological profile and quality of life of patients with oral lichen planus. J Appl Oral Sci. 2018 Jan 18;26:e20170146. doi: 10.1590/1678-7757-2017-0146. PMID 29364344
- [Background] Ramalingam S, Malathi N, Thamizhchelvan H, Sangeetha N, Rajan ST. Role of Mast Cells in Oral Lichen Planus and Oral Lichenoid Reactions. Autoimmune Dis. 2018 Jan 17;2018:7936564. doi: 10.1155/2018/7936564. eCollection 2018. PMID 29593898
- [Background] Regezi JA, Dekker NP, MacPhail LA, Lozada-Nur F, McCalmont TH. Vascular adhesion molecules in oral lichen planus. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 1996 Jun;81(6):682-90. doi: 10.1016/s1079-2104(96)80074-6. PMID 8784900
- [Background] Scott J, Huskisson EC. Graphic representation of pain. Pain. 1976 Jun;2(2):175-84. No abstract available. PMID 1026900
- [Background] Kongiel-Chablo I. [Behavior of complex cyanides in natural water with high rate of contamination]. Rocz Panstw Zakl Hig. 1966;17(1):95-102. No abstract available. Polish. PMID 5942912
- [Background] Swift JC, Rees TD, Plemons JM, Hallmon WW, Wright JC. The effectiveness of 1% pimecrolimus cream in the treatment of oral erosive lichen planus. J Periodontol. 2005 Apr;76(4):627-35. doi: 10.1902/jop.2005.76.4.627. PMID 15857105
- [Background] Thongprasom K, Luangjarmekorn L, Sererat T, Taweesap W. Relative efficacy of fluocinolone acetonide compared with triamcinolone acetonide in treatment of oral lichen planus. J Oral Pathol Med. 1992 Nov;21(10):456-8. doi: 10.1111/j.1600-0714.1992.tb00974.x. PMID 1460584
- [Background] Tripathi S, Bruch D, Kittur DS. Ginger extract inhibits LPS induced macrophage activation and function. BMC Complement Altern Med. 2008 Jan 3;8:1. doi: 10.1186/1472-6882-8-1. PMID 18173849
- [Background] Tripathi P, Tripathi P, Kashyap L, Singh V. The role of nitric oxide in inflammatory reactions. FEMS Immunol Med Microbiol. 2007 Dec;51(3):443-52. doi: 10.1111/j.1574-695X.2007.00329.x. Epub 2007 Sep 27. PMID 17903207
- [Background] van der Meij EH, van der Waal I. Lack of clinicopathologic correlation in the diagnosis of oral lichen planus based on the presently available diagnostic criteria and suggestions for modifications. J Oral Pathol Med. 2003 Oct;32(9):507-12. doi: 10.1034/j.1600-0714.2003.00125.x. PMID 12969224
- [Background] Xue JL, Fan MW, Wang SZ, Chen XM, Li Y, Wang L. A clinical study of 674 patients with oral lichen planus in China. J Oral Pathol Med. 2005 Sep;34(8):467-72. doi: 10.1111/j.1600-0714.2005.00341.x. PMID 16091113
- [Background] Yildirim B, Senguven B, Demir C. Prevalence of herpes simplex, Epstein Barr and human papilloma viruses in oral lichen planus. Med Oral Patol Oral Cir Bucal. 2011 Mar 1;16(2):e170-4. doi: 10.4317/medoral.16.e170. PMID 21196875
- [Background] Zakrzewska JM, Chan ES, Thornhill MH. A systematic review of placebo-controlled randomized clinical trials of treatments used in oral lichen planus. Br J Dermatol. 2005 Aug;153(2):336-41. doi: 10.1111/j.1365-2133.2005.06493.x. PMID 16086745
- [Background] de Wied D. [Neuropeptides and behavior. The neuropeptide concept]. Ned Tijdschr Geneeskd. 1979 Sep 15;123(37):1589-90. No abstract available. Dutch. PMID 39262
- [Background] Van Zee KJ, Coyle SM, Calvano SE, Oldenburg HS, Stiles DM, Pribble J, Catalano M, Moldawer LL, Lowry SF. Influence of IL-1 receptor blockade on the human response to endotoxemia. J Immunol. 1995 Feb 1;154(3):1499-507. PMID 7822813
- [Background] Scully C, el-Kom M. Lichen planus: review and update on pathogenesis. J Oral Pathol. 1985 Jul;14(6):431-58. doi: 10.1111/j.1600-0714.1985.tb00516.x. PMID 3926971
- [Background] Sugerman PB, Savage NW, Walsh LJ, Zhao ZZ, Zhou XJ, Khan A, Seymour GJ, Bigby M. The pathogenesis of oral lichen planus. Crit Rev Oral Biol Med. 2002;13(4):350-65. doi: 10.1177/154411130201300405. PMID 12191961
- [Background] Thongprasom K, Dhanuthai K. Steriods in the treatment of lichen planus: a review. J Oral Sci. 2008 Dec;50(4):377-85. doi: 10.2334/josnusd.50.377. PMID 19106464
- [Background] Kramer IR, Lucas RB, Pindborg JJ, Sobin LH. Definition of leukoplakia and related lesions: an aid to studies on oral precancer. Oral Surg Oral Med Oral Pathol. 1978 Oct;46(4):518-39. No abstract available. PMID 280847
- [Background] Atterhog JH, Duner H, Pernow B. Experience with pindolol, a betareceptor blocker, in the treatment of hypertension. Am J Med. 1976 May 31;60(6):872-6. doi: 10.1016/0002-9343(76)90907-4. PMID 14501
- See also: Related Info — https://www.elsevier.com/books/brenners-encyclopedia-of-genetics/maloy/978-0-12-374984-0
- See also: Related Info — https://www.jstage.jst.go.jp/article/josnusd/49/2/49_2_89/_article
- See also: Related Info — https://www.researchgate.net/publication/289537527_Efficacy_of_topical_curcumin_in_the_management_of_oral_lichen_planus_A_randomized_controlled_trial
- See also: Related Info — https://www.taylorfrancis.com/books/edit/10.1201/9781420023367/ginger-nirmal-babu-ravindran
- See also: Related Info — https://www.researchgate.net/publication/339452507_Assessment_of_Anti-inflammatory_Effect_of_Ginger_on_Mucositis_Induced_by_Cetuximab_Drug_in_Rats
- See also: Related Info — https://adjc.journals.ekb.eg/article_68490.html